CLINICAL TRIAL: NCT06860321
Title: Photodynamic Treatment in the Management of Residual Biofilm - a Crossover Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: Metropolia University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PhoBCo
Record Dates: First submitted 2025-02-26; First posted 2025-03-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults; Plaque, Dental
Keywords: aPDT; photodynamic treatment; plaque control
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Subjects are randomly divided into two group A and B. Data will be collected in two non-consecutive days to allow time for biofilm to re-form in the mouth.
  On study day 1, in both groups, teeth are cleaned at the study site by the participants themselves with an electric toothbrush and appropriate interdental cleaning tools, followed by plaque staining. The teeth are then scanned thoroughly with an oral scanner.
  Group A participants will perform a second dental cleaning themselves with an electric toothbrush and appropriate interdental cleaning tools, followed by plaque staining and scanning.
  Group B participants will perform a second dental cleaning themselves with Lumoral according to manufacture's instructions, followed by cleaning themselves with an electric toothbrush and appropriate interdental cleaning tools, followed by plaque staining and scanning.
  On study day 2, groups A and B will swap places and perform the same procedures as the other group on study day 1.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A day 1, and Group B day 2 (Active Comparator): 1) and 2) Electric toothbrushing and flossing, plaque staining and dental scan performed twice.
  Interventions: Other: Regular oral self care
- Group A day 2, and Group B day 1 (Experimental): 1. One minute of Lumorinse mouth rinse swishing followed by 10 minutes of Lumoral device use, followed by electric toothbrushing and flossing.
  2. Electric toothbrushing and flossing, plaque staining and dental scan performed twice.
  Interventions: Device: Adjunct antibacterial home-use dual-light medical device

INTERVENTIONS:
Device: Adjunct antibacterial home-use dual-light medical device — Crossover active intervention.
  Arms: Group A day 2, and Group B day 1
Other: Regular oral self care — Crossover regular intervention.
  Arms: Group A day 1, and Group B day 2

SUMMARY:
This research introduces a home-use dual-light antibacterial medical device and its possible added value as part of traditional dental self-care. The aim of the study is to investigate, using a randomized cross-over study design, whether home-use dual-light antibacterial treatment is more effective in reducing residual biofilm than mechanical, traditional cleaning of teeth and interdental spaces.

DETAILED DESCRIPTION:
The antimicrobial effect of aPDT is based on the principle that light as such activates a non-toxic, photosensitive molecule, generating reactive oxygen species that kill the bacterium. Applications of aPDT in dentistry include the treatment of bacterial and fungal infections and the diagnosis of lesions. In dental treatment, regular photodynamic treatment with dual-light has been shown to be beneficial for the gingival health of dental implants and to reduce the amount of visible plaque (VPI). Photodynamic treatment has also been shown to slow down the amount of biofilm re-forming in the mouth.

The simultaneous use of blue light and near-infrared light operating at 810 nm and 405 nm has been shown to reduce Staphylococcus aureus more effectively than using only a single light source. The use of indocyanine green as a photosensitizer in dual-light phototherapy has also been shown to be effective in eliminating Streptococcus oralis. Indocyanine green has otherwise low toxicity to dental restorative materials and to non-target host tissue. Indocyanine green is also very suitable as a photosensitizer due to its high absorption peak. Indocyanine green-mediated photodynamic therapy as an adjunct to non-surgical periodontal treatment has been shown to improve treatment outcomes for dental adhesive tissue diseases with statistically significant results at 3 months and 6 months after treatment with periodontitis patients. There is in vitro evidence for the efficacy of indocyanine green specifically against periodontal pathogens.

Tooth decay, gingivitis and periodontitis are common oral infections associated with tooth extraction and are caused by bacteria living in the mouth. In total, more than 500 different species of bacteria can be found in the mouth. The normal flora of a healthy mouth is rich in a variety of microbes that start to multiply from birth.

Bacteria of different species form biofilms, or plaques (bacterial communities), on the tooth surfaces, some of which mutate to become pro-inflammatory. Most oral diseases are multifactorial. A high-sugar diet, poor oral hygiene, general diseases, dry mouth, ill-fitting dentures or antimicrobial therapy can affect the microbial balance in the mouth and thus contribute to the development of oral diseases. Locally, oral areas are affected by possible plaque overgrowth, orthodontic appliances, open caries deposits and partially erupted wisdom teeth, which provide an easy attachment site for bacterial pathogens and a challenging area to clean.

As biofilm accumulates at the gum line over several days, it causes the tissue to release inflammatory neurotransmitters that call on defense cells from the bloodstream to destroy bacteria. Inflammation of the gums appears as swelling, redness and bleeding on cleaning. If gingivitis becomes chronic, it is a risk for periodontitis, which is the inflammation and tissue destruction of the attachment tissues. Periodontitis is manifested in the mouth as inflammation of the attachment tissues, with deepening of the gum pockets around the tooth, increased tooth mobility, and alveolar leakage on X-rays.

Careful, daily self-care and regular dental hygiene are the most important preventive measures for oral and jaw infections and dental infections. The surface of the tooth does not clean itself like the surface of the mucous membrane or skin through natural taming, so it must be cleaned mechanically. It is recommended to brush the teeth twice a day for two minutes with fluoride toothpaste and to brush the interdental spaces every 24 hours with a suitable instrument.

Lumoral® is a powerful LED light device with a mouthpiece operating blue light at 405 nm and near-infrared light at 810 nm. The Lumoral® treatment involves a combination of the use of mouth rinse inculding indocyanine green , Lumorinse®, and the Lumoral® dual-light mouthpiece. A tablet of Lumorinse® is dissolved in 30 millilitres of water to form a mouthwash, which is swished around the oral cavity for 60 seconds. After using the mouthwash, the Lu-moral® mouthpiece is placed in the mouth for 10 minutes of light activation. After use, the teeth are cleaned by brushing and cleaning the interdental spaces.

The active photosensitive substance of Lumorinse® adheres to the surface of the dental plaque, and the targeted light from the mouthpiece produces an antibacterial effect in the mouth. Lumoral® does not cause bacterial resistance, making it suitable for regular use. The treatment is bacterio-selective, meaning that it targets only harmful microbes in the mouth and does not affect the normal oral flora.

The purpose of this study is to investigate the amount of residual biofilm by comparing conventional tooth cleaning with the additional cleaning of teeth with Lumoral®. The aim is to determine whether Lumoral® treatment reduces the amount of residual biofilm in the mouth in adults in general good oral health.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent voluntarily
* Good general health

Exclusion Criteria:

* Periodontitis
* Inability to perform regular oral self-care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rustogi plaque index | 30 minutes
  The index divides the outer or inner surface of the tooth into 9 parts, based on which the amount of plaque is scored. Each tooth can score a maximum of 18 points and a minimum of 0 points at the analysis stage. The more points, the more plaque on the tooth surface is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mikko Kylmänen, Master of Health Care, Study Director — Koite Health Oy; Saila Pakarinen, Master of Arts in Education, Principal Investigator — Metropolia University of Applied Sciences
Locations (1):
- Oral Hammaslääkärit, Helsinki Bulevardi, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashir NZ, Singh HA, Virdee SS. Indocyanine green-mediated antimicrobial photodynamic therapy as an adjunct to periodontal therapy: a systematic review and meta-analysis. Clin Oral Investig. 2021 Oct;25(10):5699-5710. doi: 10.1007/s00784-021-03871-2. Epub 2021 Mar 12. PMID 33710461
- [Background] Cieplik F, Deng D, Crielaard W, Buchalla W, Hellwig E, Al-Ahmad A, Maisch T. Antimicrobial photodynamic therapy - what we know and what we don't. Crit Rev Microbiol. 2018 Sep;44(5):571-589. doi: 10.1080/1040841X.2018.1467876. Epub 2018 May 11. PMID 29749263
- [Background] Huang YY, Sharma SK, Carroll J, Hamblin MR. Biphasic dose response in low level light therapy - an update. Dose Response. 2011;9(4):602-18. doi: 10.2203/dose-response.11-009.Hamblin. Epub 2011 Sep 2. PMID 22461763
- [Background] Karu T. Primary and secondary mechanisms of action of visible to near-IR radiation on cells. J Photochem Photobiol B. 1999 Mar;49(1):1-17. doi: 10.1016/S1011-1344(98)00219-X. PMID 10365442
- [Background] Kessel D. Photodynamic Therapy: A Brief History. J Clin Med. 2019 Oct 2;8(10):1581. doi: 10.3390/jcm8101581. PMID 31581613
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Nikinmaa S, Podonyi A, Raivio P, Meurman J, Sorsa T, Rantala J, Kankuri E, Tauriainen T, Patila T. Daily Administered Dual-Light Photodynamic Therapy Provides a Sustained Antibacterial Effect on Staphylococcus aureus. Antibiotics (Basel). 2021 Oct 13;10(10):1240. doi: 10.3390/antibiotics10101240. PMID 34680821
- [Background] Pakarinen S, Saarela RKT, Valimaa H, Heikkinen AM, Kankuri E, Noponen M, Alapulli H, Tervahartiala T, Raisanen IT, Sorsa T, Patila T. Home-Applied Dual-Light Photodynamic Therapy in the Treatment of Stable Chronic Periodontitis (HOPE-CP)-Three-Month Interim Results. Dent J (Basel). 2022 Nov 2;10(11):206. doi: 10.3390/dj10110206. PMID 36354651
- [Background] Parker S. The use of diffuse laser photonic energy and indocyanine green photosensitiser as an adjunct to periodontal therapy. Br Dent J. 2013 Aug;215(4):167-71. doi: 10.1038/sj.bdj.2013.790. PMID 23969654
- [Background] Rustogi KN, Curtis JP, Volpe AR, Kemp JH, McCool JJ, Korn LR. Refinement of the Modified Navy Plaque Index to increase plaque scoring efficiency in gumline and interproximal tooth areas. J Clin Dent. 1992;3(Suppl C):C9-12. PMID 1306676
- [Background] Stajer A, Kajari S, Gajdacs M, Musah-Eroje A, Barath Z. Utility of Photodynamic Therapy in Dentistry: Current Concepts. Dent J (Basel). 2020 May 7;8(2):43. doi: 10.3390/dj8020043. PMID 32392793
- See also: Hentilä, J. et al. (2021). Dual-Light Photodynamic Therapy Effectively Eliminates Streptococcus Oralis Biofilms. JoP&PS 24. — https://journals.library.ualberta.ca/jpps/index.php/JPPS/article/view/32084
- See also: WHO. 2022. Global oral health status report: towards universal health coverage for oral health by 2030. Geneva. — https://www.who.int/publications/i/item/9789240061484